CLINICAL TRIAL: NCT00870805
Title: A Controlled Study of Ultrabrief Pulsewidth ECT (Electroconvulsive Therapy)
Brief Title: Ultrabrief Pulsewidth Electroconvulsive Therapy (ECT)
Acronym: UB ECT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of New South Wales (Other)
Collaborators: Northside Clinic, Australia (Other); The Melbourne Clinic, Australia (Unknown); St George Hospital, Australia (Other); Wandene Private Hospital, Australia (Unknown)
Responsible Party: Associate Professor Colleen Loo, University of New South Wales
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UNSW HREC 08322
Record Dates: First submitted 2009-03-26; First posted 2009-03-27 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2011-09

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- bilateral-ultrabrief ECT (Experimental): Patients will be treated with an ultrabrief (0.3ms) pulse with a bilateral placement at 3-4 times seizure threshold.
  Interventions: Procedure: bilateral ultrabrief ECT
- bilateral standard ECT (Active Comparator): Patients will be treated with a standard (1.0ms) pulse with a bilateral placement at 1.5 times seizure threshold.
  Interventions: Procedure: bilateral standard ECT
- right-unilateral ultrabrief ECT (Experimental): Patients will be treated with an ultrabrief (0.3ms) pulse with a right unilateral placement at 8 times seizure threshold.
  Interventions: Procedure: right-unilateral ultrabrief ECT
- right-unilateral standard ECT (Active Comparator): Patients will be treated with a standard (1.0ms) pulse with a right unilateral placement at 5 times seizure threshold.
  Interventions: Procedure: right-unilateral standard ECT

INTERVENTIONS:
Procedure: bilateral ultrabrief ECT — Bilateral ECT at 3-4 times seizure threshold with an ultrabrief pulse (0.3ms)
  Arms: bilateral-ultrabrief ECT
Procedure: bilateral standard ECT — Bilateral ECT with at 1.5 times seizure threshold with a standard pulse (1.0ms)
  Arms: bilateral standard ECT
Procedure: right-unilateral ultrabrief ECT — Right-unilateral ECT at 6 times seizure threshold with an ultrabrief pulse (0.3ms)
  Arms: right-unilateral ultrabrief ECT
Procedure: right-unilateral standard ECT — Right-unilateral ECT with at 5 times seizure threshold with a standard pulse (1.0ms)
  Arms: right-unilateral standard ECT

SUMMARY:
Electroconvulsive Therapy (ECT) remains essential to contemporary psychiatric practice and is one of the safest and most effective treatments available for depression. Despite modern advances in pharmacotherapy, about 15-20 per cent of all hospitalised patients receive treatment with ECT. Its use, however, is limited by concerns over associated cognitive side effects.

Recent research has suggested that using an ultrabrief pulsewidth with ECT may greatly reduce cognitive side effects, while maintaining efficacy (Sackeim et al 2008). Preliminary results were positive for unilateral ECT, however, suggest that for bilateral ECT, dosing may need to be adjusted to preserve efficacy while reducing side effects. This study will examine the relative cognitive side effects and efficacy of right unilateral and bilateral ECT given with a standard pulsewidth or an ultrabrief pulsewidth. Some participants will also receive an MRI scan before and after ECT.

ELIGIBILITY:
Inclusion Criteria:

* Subjects meet criteria for a DSM-IV-TR Major Depressive Episode
* Total MADRS score >/= 25
* Age >/= 18 years
* Educated or working in an English medium setting

Exclusion Criteria:

* Diagnosis (as defined by DSM-IV-TR) of any psychotic disorder (lifetime with exception of Major Depressive Episode with psychotic features); rapid cycling bipolar disorder, eating disorder (current or within the past year); obsessive compulsive disorder (lifetime); post-traumatic stress disorder (current or within the past year).
* history of drug or alcohol abuse or dependence (as per DSM-IV-TR) in the last 6 months (except nicotine and caffeine).
* ECT in last 3 months
* Subject requires an urgent clinical response due to inanition, psychosis or high suicide risk
* unable to give informed consent
* score < 24 on Mini Mental State Examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2009-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change in scores on Memory Tests | Before ECT, after 6 ECT treatments, after final ECT treatment, one month and six month follow-up

SECONDARY OUTCOMES:
Change in scores on Depression Rating Scale | Before ECT, after each week of treatment, at the end of the ECT course

CONTACTS AND LOCATIONS:
Overall Officials: Assoc/Prof Colleen K Loo, MBBS, FRANZCP, MD, Principal Investigator — University of New South Wales; Prof Isaac Schweitzer, MBBS, FRANZCP, MD, Principal Investigator — The Melbourne Clinic
Locations (3):
- Australia (3):
  - St George Hospital, Kogarah, New South Wales
  - Wandene Private Hospital, Kogarah, New South Wales
  - The Melbourne Clinic, Melbourne, Victoria

REFERENCES:
- [Background] Loo CK, Schweitzer I, Pratt C. Recent advances in optimizing electroconvulsive therapy. Aust N Z J Psychiatry. 2006 Aug;40(8):632-8. doi: 10.1080/j.1440-1614.2006.01862.x. PMID 16866758
- [Background] Loo C, Sheehan P, Pigot M, Lyndon W. A report on mood and cognitive outcomes with right unilateral ultrabrief pulsewidth (0.3 ms) ECT and retrospective comparison with standard pulsewidth right unilateral ECT. J Affect Disord. 2007 Nov;103(1-3):277-81. doi: 10.1016/j.jad.2007.06.012. Epub 2007 Aug 16. PMID 17706790
- [Background] Loo CK, Sainsbury K, Sheehan P, Lyndon B. A comparison of RUL ultrabrief pulse (0.3 ms) ECT and standard RUL ECT. Int J Neuropsychopharmacol. 2008 Nov;11(7):883-90. doi: 10.1017/S1461145708009292. Epub 2008 Aug 28. PMID 18752719
- [Background] Sackeim HA, Prudic J, Nobler MS, Fitzsimons L, Lisanby SH, Payne N, Berman RM, Brakemeier EL, Perera T, Devanand DP. Effects of pulse width and electrode placement on the efficacy and cognitive effects of electroconvulsive therapy. Brain Stimul. 2008 Apr;1(2):71-83. doi: 10.1016/j.brs.2008.03.001. PMID 19756236
- [Background] Sienaert, P., Vansteelandt, K., Demyttenaere, K., & Peuskens, J. (2006). Comparison of bifrontal and unilateral ultra-brief pulse electroconvulsive therapy for depression. European Neuropsychopharmacology, 16 (suppl 4), S28.
- [Derived] Martin D, Katalinic N, Hadzi-Pavlovic D, Ingram A, Ingram N, Simpson B, McGoldrick J, Dowling N, Loo C. Cognitive effects of brief and ultrabrief pulse bitemporal electroconvulsive therapy: a randomised controlled proof-of-concept trial. Psychol Med. 2020 May;50(7):1121-1128. doi: 10.1017/S0033291719000989. Epub 2019 May 2. PMID 31056081
- [Derived] Loo CK, Katalinic N, Smith DJ, Ingram A, Dowling N, Martin D, Addison K, Hadzi-Pavlovic D, Simpson B, Schweitzer I. A randomized controlled trial of brief and ultrabrief pulse right unilateral electroconvulsive therapy. Int J Neuropsychopharmacol. 2014 Dec 5;18(1):pyu045. doi: 10.1093/ijnp/pyu045. PMID 25522389